CLINICAL TRIAL: NCT02630433
Title: Randomised Controlled Trial of Index Cholecystectomy Versus Scheduled Cholecystectomy in Biliary Pancreatitis
Brief Title: Trial of Index Cholecystectomy Versus Scheduled Cholecystectomy in Biliary Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Gabriel Sandblom, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Gallstenspancreatitistudien
Record Dates: First submitted 2015-12-06; First posted 2015-12-15 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Pancreatitis
Keywords: Biliary pancreatitis; Cholecystectomy
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Index cholecystectomy (Experimental): Cholecystectomy within 48 hours after inclusion.
  Interventions: Procedure: Index cholecystectomy
- Scheduled cholecystectomy (Active Comparator): Cholecystectomy 6 weeks after inclusion.
  Interventions: Procedure: Scheduled cholecystectomy

INTERVENTIONS:
Procedure: Index cholecystectomy — Cholecystectomy performed within 48 hours after inclusion, before discharge after admission for acute biliary pancreatitis.
  Arms: Index cholecystectomy
Procedure: Scheduled cholecystectomy — Cholecystectomy performed as a scheduled procedure 6 weeks after the first admission.
  Arms: Scheduled cholecystectomy

SUMMARY:
There are controversies optimal timing for cholecystectomy in patients with mild biliary pancreatitis. The safety of cholecystectomy performed during an episode of pancreatitis has been questioned. The aim of the present randomized controlled trial is to compare the outcome in terms of recurrent pancreatitis and gallstone-related events between index cholecystectomy, performed during the first admission for acute pancreatitis, and scheduled cholecystectomy, performed 4-6 weeks after discharge.

DETAILED DESCRIPTION:
Background:

There is still considerable debate regarding the optimal timing of cholecystectomy in mild biliary pancreatitis. It is widely accepted to wait until the patient's clinical condition allows performing cholecystectomy in severe biliary pancreatitis with systemic or local complications. On the other hand, the recommendations are not very clear when it comes to patients with mild biliary pancreatitis. The British Society of Gastroenterology and American Gastroenterological Association guidelines recommendation is to perform cholecystectomy within 2-to 4- week interval after the initial episode. However, the safety of cholecystectomy performed during an episode of pancreatitis is also controversial.

In a systematic review the overall readmission rate was 18% after index cholecystectomy, 8% for recurrent biliary pancreatitis, 3 % for acute cholecystitis and 7 % for biliary colic.

Methods The study is performed as a Randomised controlled trials with two parallel arms and a ratio of 1:1. Patients admitted with acute pancreatitis are checked for eligibility criteria for the study. Mild pancreatitis is defined as pancreatitis without local complications such as necrosis or organ failure. Patients who are eligible obtained oral and written information about the study and invited to be included. Patients who accept participation sign a consent form and are included. The included patients are randomized into index cholecystectomy (IC) or scheduled cholecystectomy (SC).

Randomization is done with a sealed envelope system. The allocation sequence is created by an online random generator. There is no blocking. After randomization, the patient as well as the responsible are immediately informed about the allocation.

The IC and SC are protocolled to be performed within 24-48 hours from randomization, and after 6 weeks from discharge respectively. Daily blood samples, pain and well-being scores are obtained during index admission until discharge, at 1-month follow-up for SC group and at the scheduled cholecystectomy. Quality of life is assessed with SF-36 prior to randomization and 4 weeks after inclusion. Pain is measured with the McGill Pain Questionnaire before randomization and daily until discharge of two days after inclusion.

Sample size estimation If IC reduces the risk of gallstone- or treatment-related adverse events from 40% to 10%, a total sample of 32 patients in each group is required in order to reach a chance of 80% of detecting a significant difference at the p<0.05 level. In order to compensate of drop-outs, a total sample of 70 is stipulated.

ELIGIBILITY:
Inclusion Criteria:

* S-Amylase >3 microkat/L
* One or more gallstones with diameter < 2 cm
* S-CRP < 150 mg/L the first 24 hours

Exclusion Criteria:

* Multiple organ failure
* Solitary gallstone with diameter >2 cm
* Concurrent cholangitis
* Hospital stay exceeding 72 hours before screening for inclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-08; Primary Completion 2017-11-12 (Actual); Study Completion 2017-11-12 (Actual)

PRIMARY OUTCOMES:
Recurrent acute pancreatitis | 6 weeks
  Relapse of acute pancreatitis in the scheduled cholecystectomy arm

SECONDARY OUTCOMES:
Complications related to the cholecystectomy | 30 days
  Complications according to the Clavien-Dindo classification
Markers of inflammatory activity | 3 days
  Inflammatory response measured with CRP and interleukins
Health-related quality of life measured with SF-36 | 6 weeks
  Health-related quality of life measured with SF-36 the day of inclusion and 6 weeks after inclusion
Cost-effectiveness | 6 weeks
  Costs from hospital stay, the surgical procedure and sick leave.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Sandblom, Ass prof, Principal Investigator — Karolinska Institutet, CLINTEC
Locations (1):
- Karolinska University Hospital, Center for Digestive Diseases, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Noel R, Arnelo U, Lundell L, Hammarqvist F, Jumaa H, Enochsson L, Sandblom G. Index versus delayed cholecystectomy in mild gallstone pancreatitis: results of a randomized controlled trial. HPB (Oxford). 2018 Oct;20(10):932-938. doi: 10.1016/j.hpb.2018.03.016. Epub 2018 Apr 25. PMID 29703649